CLINICAL TRIAL: NCT00676013
Title: The Use of Alloderm and Other Skin Substitutes in Acute Burn Treatment and Burn Scar Reconstruction
Brief Title: Comparison of Skin Substitutes Used in Burn Care
Acronym: Quad
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to continue study following Hurricane Ike.
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 97-286
Record Dates: First submitted 2007-12-26; First posted 2008-05-12 (Estimated); Results first posted 2019-12-16 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2018-08

CONDITIONS: Burns
Keywords: Burns; Skin grafting; AlloDerm; Integra; Homograft; Autograft; Burn Scar
MeSH Terms: conditions — Burns | interventions — integra artificial skin; Alloderm; Transplantation, Homologous; Transplantation, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alloderm, Integra, Homograft, Autograft (Experimental): Burn debridement and grafting using interventions of 1) AlloDerm, 2) Integra, 3) Homograft and 4) Autograft on four separate sites on each patient
  Interventions: Procedure: Integra; Procedure: AlloDerm; Procedure: Homograft; Procedure: Autograft

INTERVENTIONS:
Procedure: Integra — Grafting using the Commercial product Integra as a skin substitute over full thickness burn following excision.
  Other Names: Artificial dermis
Procedure: AlloDerm — Grafting using the commercial product AlloDerm as a skin substitute
  Other Names: Cadaver skin
Procedure: Homograft — Grafting using homograft as a skin substitute
  Other Names: Cadaver Skin
Procedure: Autograft — grafting using patients own skin from a separate donor site

SUMMARY:
The purpose of this study is to determine if using a DERMAL LAYER under skin grafts:

1. will reduce scar formation of skin grafts
2. will reduce burn wound contractures
3. will improve functional outcome of joints requiring grafts

Compare scarring outcome of Dermal products

DETAILED DESCRIPTION:
Various skin substitutes are compared for healing, scar and functional and cosmetic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Burn injury requiring grafting
* 0 years-90 years

Exclusion Criteria:

* Partial thickness burns only

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 1997-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David N Herndon, MD, Principal Investigator — University of Texas
Locations (2):
- United States (2):
  - University of Texas Medical Branch, Galveston, Galveston, Texas
  - University of Texas Medical Branch, Galveston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the Galveston Burn Unit following an acute burn injury that were diagnosed with 3rd degree burns. Study was active between 1997-2011.
Pre-assignment Details: Patients were enrolled before their surgical procedure. After consent was obtained. After the surgical site was identified, the site was randomized to receive the various skin products.
Groups:
- Alloderm, Integra, Homograft, Autograft: Grafting with alloderm, Integra, Homograft, and/or Autograft on each patient. Different sites were then compared.
Period: Overall Study
Arm/Group | Alloderm, Integra, Homograft, Autograft
Started | 158
Completed | 157
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Alloderm, Integra, Homograft, and/or Autograft: Grafting with alloderm, integra, homograft and/or autograft. Various treatment sites were then compared.
Arm/Group | Alloderm, Integra, Homograft, and/or Autograft
Number analyzed (Participants) | 158
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 158
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 110
Region of Enrollment [Number; unit: participants]
  United States | 158

OUTCOME MEASURES:

1. Primary Outcome: Burn Scar Comparison
Description: Burn scar is measured scar using the Vancouver Scar Scale (range 0-12) for each of the various skin substitutes used in grafting. Vancouver Scar Scale measure burn scarring assessing categories of redness/vascularity, hardness, pigmentation and scar height. Each item has a scale of 0-3. Score for each category is summed together for a total score between 0-12. The total score is generally used in the burn community, therefore the total score will be reported. Lower scores are better; higher scores are worse.
Time Frame: 2 years post burn injury
Population: Each site grafted with a skin substitute was analyzed with a Scar Assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- AlloDerm: Surgery using alloDerm. Various treatment sites were then compared.
- Integra: Surgery with Integra grafting followed with autografting
- Homograft: Surgery using Homograft followed with autografting
- Autograft: Surgery with Autografting
Arm/Group | AlloDerm | Integra | Homograft | Autograft
Number analyzed (Participants) | 158 | 158 | 158 | 158
units on a scale
  Scar Score 6 months post burn | 10.7 (1.0) | 6.9 (1.4) | 12.0 (1.8) | 11.6 (.8)
  Scar Score 24 months post burn | 5.7 (.9) | 4.7 (.8) | 4.8 (.7) | 5.6 (.8)
Statistical Analysis 1: Comparison: AlloDerm vs Integra vs Homograft vs Autograft; We conducted a multiple four group comparison (all pairwise comparisons were conducted). An Anova was conducted to assess statistical significance; Test type: Other — ANOVA and all pairwise comparisons using Tukey test; p = 0.05, ANOVA — 0.05 is a threshold for statistical significance; Multiple pairwise comparisons = 0.05; 0.05

ADVERSE EVENTS:
Time Frame: 1997-2011
Groups:
- AlloDerm, Integra, Homograft, Autograft: Skin product used on each of the four test sites on each patient
Arm/Group | AlloDerm, Integra, Homograft, Autograft
Serious Adverse Events (participants affected / at risk) | 9/158
Other Adverse Events (participants affected / at risk) | 3/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AlloDerm, Integra, Homograft, Autograft (N=158)
Aspiration and Death (Respiratory, thoracic and mediastinal disorders) | 1 (1) — 2001: Following discharge from hospital, patient aspirated while sleeping. Advanced Cardiac Life Support provided however patient expired. PI felt Adverse Event not related to study.
Invasive infection and death (Infections and infestations) | 1 (1) — 2001: 74% burn admitted with invasive infection. Developed multi organ failure,, coded and expired. Patient never started study. PI stated Adverse Event not related to study.
90% burn admitted with renal failure, died (Renal and urinary disorders) | 1 (1) — 2001: 90% burn admitted with renal failure. After most of burns were grafted, renal failure worsened, patient eventually died. PI stated unlikely related to study.
leg ischemia (Vascular disorders) | 1 (1) — 2001: Arterial line placed for surgical procedure, right leg became ischemic. Treated with anticoagulants. No long term complications. PI stated not related to study.
Invasive infection, Multi organ failure, death (Infections and infestations) | 1 (1) — 2001: 85% burn patient admitted with invasive infection. Developed sepsis, renal failure, multi organ failure. Patient allowed to die.
Respiratory status compromised (Respiratory, thoracic and mediastinal disorders) | 2 (2) — 2001: Chest tube pulled out. PI stated not related to study. 2001: Plugged Endotracheal tube x2. Endotracheal Tube pulled and replaced. PI opinion is Adverse Event is not related to study.
hypoglycemia (Endocrine disorders) | 2 (2) — 2001 Patient on insulin drip, glucose decreased to 35. Glucose treated,Insulin stopped. PI opinion:not related to study. 2001: Patient on insulin drip. Glucose decreased to 30. Patient treated, insulin stopped. PI opinion:not related to study.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AlloDerm, Integra, Homograft, Autograft (N=158)
Hematoma (Vascular disorders) | 2 (2) — 2003: Hematoma following femoral IV line placement. PI opinion is Adverse Event is not related to study. 2006: hematoma developed following femoral IV line placement. PI opinion is Adverse Event is not related to study.
Fall and open wound (Skin and subcutaneous tissue disorders) | 1 (1) — 2001: Patient fell trying to push chair and ripped skin open.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No